CLINICAL TRIAL: NCT04289363
Title: Emergency Department Outcomes for Patients With Opioid Use Disorder
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-01444; 3UG1DA013035-18S3 (NIH)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ED patients: Administrative and health record data will be examined to assess rates of screening, assessment, eligibility determination, etc.
  Interventions: Behavioral: Clinical program implementation

INTERVENTIONS:
Behavioral: Clinical program implementation — Using mixed methods and triangulating multiple sources of data collected over the course of parent and ancillary studies to evaluate the feasibility, acceptability, sustainability, and impact of the ED-initiated BUP clinical program and implementation facilitation strategy and identify factors influencing diffusion and effectiveness. Converging provider and patient perspectives and field notes with process measures and intervention outcomes, including proportions screened, treated, and engaged in treatment, will provide explanation to contextualize and better understand feasibility, acceptability, and factors associated with the rate with which the ED-initiated BUP innovation is adopted and how well it is sustained.

SUMMARY:
Using mixed methods and triangulating multiples sources of data collected over the course of the parent (CTN-0079 - NCT03544112) and the ancillary studies to evaluate the feasibility, acceptability, sustainability and impact of the emergency department (ED)-initiated Buprenorphine (BUP) clinical program and implementation facilitation strategy and identify factors influencing diffusion and effectiveness.

DETAILED DESCRIPTION:
The ancillary study will use mixed-methods combining quantitative and qualitative inquiry (interview/focus group and field notes) with administrative and health record data with some analyses including data collected from the parent CTN-0079 (NCT03544112) study. Further, qualitative data will be analyzed in the context of themes derived from CTN-0069 (NCT03023930) and CTN-0079. CTN-0079-A1 is planned to be conducted at two of the three sites of the parent study: (1) Catholic Medical Center, Manchester, New Hampshire; (2) Bellevue/NYU Health and Hospitals, New York, NY. Many of the methods, operating procedures, measures and forms will be retained or adapted from the parent study. However, CTN-0079-A1 is a new study in which lessons learned through the parent study have informed important design modifications necessary to improve study rigor and utility.

As in the parent study, CTN-0079, all clinical care (BUP and referral) will be delivered as part of each facility's clinical protocol, rather than as a research procedure. Implementation Facilitation (IF) activities will continue during ancillary trial preparation with a more intensive booster of IF activities occurring in the last month prior to trial commencement. Thereafter, all study IF support will cease and ancillary study data collection will begin. Data collection will occur over a course of approximately 12 months, divided into two 6-month study periods - the Post-IF and Maintenance Periods. A period of at least 6 months should separate the beginning of the Maintenance Period from the time of last study intervention.

ELIGIBILITY:
Inclusion Criteria:

Qualitative Population:

* Key stakeholder or opinion leader for ED-initiated BUP
* 18 years of age or older

Full Study Population & Limited Study Population:

* Be able to speak English sufficiently to understand study procedures
* Be a potential candidate for ED-initiated BUP by meeting either of the 2 criteria:

  1. Clinical determination: patient is a willing and eligible candidate for ED-initiated BUP or for whom this can be reasonably inferred, including any patient who is administered and/or prescribed BUP as part of the index ED visit.
  2. Research determination: Both a and b below must be true at the time of study enrollment:

  a) Assessment conducted by an RA indicates that the patient- (all must be true): i. has had nonmedical opioid use within the last 7 days, ii. meets DSM-5 criteria for moderate or severe opioid use disorder (OUD), iii. denies methadone use within 72 hours of ED visit registration, iv. is not engaged in formal medications for opioid use disorder (MOUD) treatment, v. is not prescribed opioids for chronic pain management, vi. reports being interested or "not sure" if interested in receiving BUP as elicited on the ED Health Survey during the index ED visit.

  b) Absence of clinical documentation associated with the ED visit indicating that the patient is not a candidate for ED-initiated BUP.

Exclusion Criteria:

Qualitative Population:

* Unwilling or unable to provide consent
* currently in jail, prison, or any inpatient overnight facility

Full Study Population:

* Unwilling or unable to provide written/electronic informed consent
* Currently engaged in formal MOUD treatment at the time of index ED visit
* Currently in jail, prison or any inpatient overnight facility as required by court of law
* Previous participation as a patient- participant in CTN-0079 or previous participation as a Full Study participant in the current study
* Presents from a medical-based extended care facility
* Current research participant in a substance use intervention study
* Inadequate locator information (unable or unwilling to provide 2 unique means of contact)
* Unable or unwilling to complete research visits at baseline and Day 30.

Limited Study Population:

* Unwilling or unable to provide written/electronic informed consent
* Currently engaged in formal MOUD treatment at the time of index ED visit
* Currently in jail, prison or any inpatient overnight facility as required by court of law
* Previous participation in the current study as a Limited study or Full study participant
* Presents from a medical-based extended care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include ED patients.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan McCormack, MD, MS, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Catholic Medical Center, Manchester, New Hampshire
  - Bellevue Hospital Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol
Time Frame: Data sets for CTN protocols will be available after (1) the primary paper has been accepted for publication, or (2) the data is locked for more than 18 months, whichever comes first.
Access Criteria: Anyone who wishes to access the data.Any purpose. Data are available indefinitely at https://datashare.nida.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Certain Outcome Measures of the current study were pre-specified to utilize participants not enrolled in the study. These participants are represented in the "Patients Identified via Chart Review" arm. As these participants were not enrolled in the study, they are not counted in the Protocol Enrollment. Enrolled participants are represented in the "ED Patients" arm.
Groups:
- Patients Identified Via Chart Review: Patients who were identified via retrospective chart review for the purpose of outcome measure analysis.
Period: Overall Study
Arm/Group | ED Patients | Patients Identified Via Chart Review
Started | 53 | 1489
Completed | 39 | 1489
Not Completed | 14 | 0
Not completed — Lost to Follow-up | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Identified Via Chart Review: Patients who were identified via chart review.
- Total: Total of all reporting groups
Arm/Group | ED Patients | Patients Identified Via Chart Review | Total
Number analyzed (Participants) | 39 | 1489 | 1528
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (10.72) | 41.3 (11.91) | 42.25 (11.315)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not all participants in the "Patients identified via Chart Review" arm had baseline Sex data collected. Thus, the total number of participants analyzed for each of these sections is less than the overall number of baseline participants.
  Participants
    number analyzed (Participants) | 39 | 1488 | 1527
    Female | 10 | 277 | 287
    Male | 29 | 1211 | 1240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Not all participants in the "Patients identified via Chart Review" arm had baseline ethnicity data collected. Thus, the total number of participants analyzed for each of these sections is less than the overall number of baseline participants.
  Participants
    number analyzed (Participants) | 39 | 1289 | 1328
    Hispanic or Latino | 7 | 198 | 205
    Not Hispanic or Latino | 32 | 1044 | 1076
    Unknown or Not Reported | 0 | 47 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Not all participants in the "Patients identified via Chart Review" arm had baseline race data collected. Thus, the total number of participants analyzed for each of these sections is less than the overall number of baseline participants.
  Participants
    number analyzed (Participants) | 39 | 1075 | 1114
    American Indian or Alaska Native | 0 | 10 | 10
    Asian | 0 | 4 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 8 | 317 | 325
    White | 27 | 658 | 685
    More than one race | 0 | 35 | 35
    Unknown or Not Reported | 4 | 50 | 54
Region of Enrollment [Number; unit: participants]
  United States | 39 | 1489 | 1528

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Received Emergency Department (ED)-Initiated/Expedited Buprenorphine (BUP)
Description: The outcome will be calculated using the following formula: [(Candidates who receive ED-initiated BUP with any disposition) + (Candidates who receive ED-expedited BUP and who are discharged)] / [(Candidates who are discharged) + (Candidates who receive ED-initiated BUP that are not discharged)].
Time Frame: Up to Month 12
Population: The overall number of participants analyzed for this outcome measure (n=1489) represents individuals identified via retrospective chart review and data matching for all adult emergency department (ED) patients identified to have nonmedical opioid use presenting to the ED during the IF, Post-IF or Maintenance periods. This outcome was not assessed among participants in the ED patients arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patients Identified Via Chart Review
Number analyzed (Participants) | 1489
Percentage of participants | 39.40 [36.7 to 42.0]

2. Primary Outcome: Percent of Participants Who Received ED-Initiated/Expedited BUP Who Were Confirmed to be Engaged in Formal Addiction Treatment for Opioid Use Disorder (OUD) on the 30th Day Following Discharge
Description: The outcome will be calculated using the following formula: (participants who are confirmed to be engaged in formal addiction treatment for Opioid Use Disorder (OUD) on the 30th day following discharge / total number of participants who received ED-initiated/expedited BUP).
Time Frame: Day 30 Post-Discharge (Up to Month 12)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ED Patients
Number analyzed (Participants) | 38
Percentage of participants | 48.3 [33.2 to 63.5]

3. Secondary Outcome: Percent of Discharged Participants Who Received ED-Initiated BUP
Description: The outcome will be calculated using the following formula: [(ED-initiated, discharged) + (ED-expedited, discharged)] / All candidates who were discharged
Time Frame: Up to Month 12
Population: The overall number of participants analyzed for this outcome measure (n=1281) represents individuals identified via retrospective chart review and data matching for all adult emergency department (ED) patients identified to have nonmedical opioid use presenting to the ED during the IF, Post-IF or Maintenance periods. This outcome was not assessed among participants in the ED patients arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patients Identified Via Chart Review
Number analyzed (Participants) | 1281
Percentage of participants | 32.10 [29.1 to 35.0]

4. Secondary Outcome: Percent of Not-Admitted Participants Who Received ED-Initiated BUP
Description: The outcome will be calculated using the following formula: (ED-initiated, not admitted) /All candidates who were not admitted
Time Frame: Up to Month 12
Population: The overall number of participants analyzed for this outcome measure (n=1317) represents individuals identified via retrospective chart review and data matching for all adult emergency department (ED) patients identified to have nonmedical opioid use presenting to the ED during the IF, Post-IF or Maintenance periods. This outcome was not assessed among participants in the ED patients arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patients Identified Via Chart Review
Number analyzed (Participants) | 1317
Percentage of participants | 28.10 [25.3 to 30.9]

5. Secondary Outcome: Percent of Participants Who Received ED-Initiated BUP
Description: The outcome will be calculated using the following formula: (ED-initiated, all) / [All discharged candidates + (ED-initiated, not discharged)]
Time Frame: Up to Month 12
Population: The overall number of participants analyzed for this outcome measure (n=1310) represents individuals identified via retrospective chart review and data matching for all adult emergency department (ED) patients identified to have nonmedical opioid use presenting to the ED during the IF, Post-IF or Maintenance periods. This outcome was not assessed among participants in the ED patients arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patients Identified Via Chart Review
Number analyzed (Participants) | 1310
Percentage of participants | 30.7 [27.8 to 33.5]

6. Secondary Outcome: Percent of Participants Who Received ED-Initiated/Expedited BUP
Description: The outcome will be calculated using the following formula: (ED-initiated/expedited, all) / [All discharged candidates + (ED-initiated/expedited, not discharged)]
Time Frame: Up to Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Patients Identified Via Chart Review
Number analyzed (Participants) | 1489
Percentage of participants | 25.4 [22.9 to 27.9]

7. Secondary Outcome: Change in Number of Days of Opioid and/or Other Drug Use as Assessed by Timeline Followback (TLFB) Assessment
Description: The TLFB assessment will elicit the participant's self-reported use of illicit substances over the previous 7 days. At the Day 30 follow-up visit the assessment period will be the 7 days preceding the Day 30 post index ED visit.
Time Frame: Baseline, Day 30
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | ED Patients
Number analyzed (Participants) | 30
Days | -2.3 [-3.7 to -0.9]

8. Secondary Outcome: Change in Number of Self-Reported Opioid-Related Overdose Events
Description: Participants will be asked to report the number of opioid-related overdose events experienced in the past 30 days through a self-report form.
Time Frame: Baseline, Day 30
Measure: Mean (95% Confidence Interval); unit: Overdose events
Arm/Group | ED Patients
Number analyzed (Participants) | 30
Overdose events | 1.78 [0.44 to 7.24]

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Among enrolled patients (participants in the ED Patients arm), serious adverse events and other (non-serious) adverse events were not assessed; only death was assessed. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not intended to be monitored/assessed among patients identified via chart review.
Arm/Group | ED Patients | Patients Identified Via Chart Review
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT04289363/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT04289363/ICF_001.pdf